CLINICAL TRIAL: NCT06927271
Title: Effectiveness, Cost-effectiveness, and Acceptability of Phone Call and Video-based Interventions to Improve Adherence to Antihypertensive Medications
Brief Title: Effectiveness of Phone Call and Video-based Interventions to Improve Adherence to Medications in Hypertensive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ghana (Other)
Responsible Party: Principal Investigator, GRACE ADJEI OKAI, Principal Investigator, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GHS-ERC:001/10/23
Record Dates: First submitted 2025-01-17; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Hypertension (Without Type 2 Diabetes Mellitus)
Keywords: hypertension; adherence; medications; mHealth; mobile technology
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the video-group (Active Comparator): In this arm, participants with uncontrolled blood pressure will receive videos via WhatsApp to educate them about the condition hypertension, side effects of medications and also remind them to take their medications. The intervention will be administered on days and time convenient for the patient and will be administered thrice weekly for 3 months. Participants in this group will receive the video intervention in addition to usual care (which is the care they receive from health facilities)
  Interventions: Other: Video based intervention
- the phone call group (Active Comparator): In this arm, participants with uncontrolled blood pressure will receive phone calls to educate them about the condition hypertension, side effects of medications and also remind them to take their medications. The intervention will be administered on days and time convenient for the patient and will be administered thrice weekly for 3 months. Participants in this group will receive the phone call intervention in addition to usual care (which is the care they receive from health facilities)
  Interventions: Other: phone call based intervention
- control group (Placebo Comparator): This group will neither receive phone call or videos. The group will only receive a message that indicates that they are being enrolled into the study.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: phone call based intervention — The phone call based intervention seek to educate patients about hypertension and the medications used. It also seeks to remind patients to take their medications. This will be done thrice weekly
  Arms: the phone call group
Other: Video based intervention — The video based intervention seek to educate patients about hypertension and the medications used. It also seeks to remind patients to take their medications. This will be done thrice weekly
  Arms: the video-group
Other: Usual Care — The usual care concerns the care the participants receive from the health facility. Participants in this group would neither receive the phonecall or video based interventions.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to find out if phone call and video-based interventions that seek to educate people with uncontrolled high blood pressure and also remind them to take their medicines will improve adherence to their medicines. It will also examine if the interventions are economical to implement. The main objectives of the study are:

* Design videos and phone call-based interventions for people with hypertension.
* Examine the effect of videos and phone call-based intervention on adherence to medication in people with hypertension.
* Calculate the costs associated with the mobile health intervention
* Examine the factors influencing acceptance of video and phone calls based interventions for improving adherence to antihypertensive medications among patients

Participants will:

* Receive the intervention thrice weekly for 3 months
* Visit the health facility at the end of 3 months for check up and measurement of outcome variables (adherence and blood pressure). Additionally, at the end of 3 months, the acceptability of the interventions will be measured among the participants who received either phone call or video.

Researchers will compare the two groups (one group will utilize phone call whereas the other videos) with the control group to see if the mobile interventions improve adherence to medicines. Only adults 18 years and above in selected health facilities in the Eastern will participate in the study. The selected participants should have uncontrolled blood pressure based on readings from last 2 visits. To be included in the study, the participants need to own a smartphone.

DETAILED DESCRIPTION:
Hypertension prevalence in adults ranges between 19 percent and 55 percent in Ghana (Agongo et al., 2020). About half of the patients diagnosed with hypertension in Ghana exhibit signs of organ damage which occur as a result of poor control of blood pressure and late detection by the health system (Atibila et al., 2021). Despite the availability of effective treatment regimen and evidence of benefits of treatment, hypertension remains poorly controlled in Ghana as studies have reported control rates ranging from 24 percent to 42 percent (Sanuade et al., 2018).

The high prevalence of uncontrolled blood pressure has been attributed mainly to poor medication adherence (Boima et al., 2015). A study conducted by Abeasi et al. (2022) in the Upper East region indicated that about 60 percent of hypertensive patients were nonadherent to their medications. Also, another study (Adomako et al., 2021) reported non-adherence rates of 49 percent and 53 percent in two hospitals in the Ashanti region. These high rates of nonadherence thwart the efforts to control and manage hypertension.

With the increase in availability and uptake of mobile phones worldwide, mobile health technologies (mHealth) have been identified as promising strategies that can be used to remind, motivate and educate patients about their disease as well as medications to improve adherence to medications in patients with hypertension (Anglada-Martinez et al., 2015; Xiong et al., 2018). Ghana has the highest mobile penetration rate in Africa (Global System for Mobile Communications Association (GSMA), 2020) and as of 2021, there were over 40 million mobile connections in the country (Kemp, 2021). The widespread use of mobile phones provides a unique opportunity for clinicians to leverage mHealth to improve medication adherence as they are incorporated widely into daily life.

Studies that have utilized mHealth interventions to improve adherence to antihypertensive medications have mostly employed short message service (SMS)(Buis et al., 2017; Leon et al., 2015; Maslakpak & Safaie, 2016; Sartori et al., 2020; Varleta et al., 2017). The challenge with text messaging or SMS is that it is difficult to apply to every context, especially in Africa where the literacy level is reported to be low (Gee et al., 2015). Also, evidence suggests that individuals with lower levels of education may not open and read the messages (Saleh et al., 2018). There is also the likelihood that people may read the messages and may not understand them (Sartori et al., 2020). Additionally, text messaging restricts the number of characters that can be sent and hence, messages sent may lack details which makes them difficult to be understood (Schoenthaler et al., 2020). Other authors have noted that the content of the messages may become monotonous resulting in message fatigue and possible withdrawal from the study (Finitsis et al., 2014; Horner et al., 2017).

Other equally important alternatives such as phone calls and videos can overcome most of the challenges associated with SMS (Asante et al., 2020; Stanczyk et al., 2016). Existing evidence from the healthcare literature suggests that videos perform better than written words since words cannot convey facial expressions and body language (Schooley et al., 2015). Again the use of videos is useful for individuals who have less education, health literacy and motivation to take medicines as it does not necessitate extensive reading of numerous pages of written material (Ben-Zeev et al., 2018). The use of phone call based interventions also increases patients confidence in the information provided and allows them to receive immediate feedback on queries about their illness or medications (Son et al., 2020). There is a paucity of studies on use of phone call and video-based interventions in improving adherence to medications in hypertensive patients in the mHealth literature (Chun-Yun Kang, 2022).

Further, most mHealth studies have focused mostly on the design and implementation of the interventions as well as examining the effectiveness of the interventions. However, it is important to understand the costs incurred for the effectiveness achieved to ascertain value of investing in the technology (Hamine et al., 2015; Rehman et al., 2017; Varleta et al., 2017). Data on the cost-effectiveness of mHealth interventions are predominantly unavailable in developing countries (Majumdar et al., 2015; Stephani et al., 2016). The economic evaluation of mobile health interventions is imperative as it helps policymakers to make decisions that ensure better resource allocation.

In Ghana, a dearth of literature exists on randomized controlled trials examining the effectiveness of mobile health interventions in improving treatment adherence in hypertensive patients. Existing studies have focused on examining the usage of smartphone applications to improve blood pressure control among stroke patients (Sarfo et al., 2019) and barriers, facilitators as well as recommended mHealth strategies to manage hypertension in patients who have recovered from stroke (Nichols et al., 2017). None of these studies considered the general hypertensive patients who can escape the possibility of experiencing stroke when they adhere to their medications and also, none utilized phone calls and video-based interventions.

Additionally, most of the mHealth studies conclude with evaluation of effectiveness of the interventions without exploring the reasons behind the results. Nonetheless, it is important to understand why the intervention is effective or not to guide future intervention development and also possible scale-up. In the context of technology, the effectiveness is likely dependent on the acceptability of the intervention by the target population which influences usage (AlSwayied et al., 2022; Sekhon et al., 2017). Very little is known about the acceptability and determinants of acceptance of mHealth interventions for the management of chronic non-communicable diseases including hypertension in developing countries (Déglise et al., 2012; Majumdar et al., 2015).

This study aims to fill the gaps in the literature by examining the effectiveness, cost-effectiveness and acceptability of video and phone call interventions in improving adherence to antihypertensive medications in Ghana using a randomized controlled trial.

Specifically, the study seeks to:

I. Design videos and phone calls-based interventions for hypertensive patients. II. Examine the effect of videos and phone call-based intervention on adherence to medication in hypertensive patients.

III. Examine the cost-effectiveness of phone call and video-based interventions in improving adherence to medications in hypertensive patients IV. Examine the factors influencing acceptance of video and phone calls-based interventions for improving adherence to antihypertensive medications among patients.

Research Questions I. Do phone calls and video-based interventions improve adherence to antihypertensive medications? II. What is the cost-effectiveness of mobile health interventions (phone calls and videos) in improving adherence to antihypertensive medications?

III. What are the factors influencing the acceptance of video and phone calls-based interventions to improve adherence to medications in hypertensive patients?

Study Design A three-armed parallel cluster randomized controlled trial (RCT) design will be utilized for the study with participants recruited from health facilities. One group will be randomized to receive phone calls in addition to care as usual. The second group will receive videos as well as usual care whereas the control group will receive usual care only. Randomisation by health facilities is chosen to evade potential contamination that could result when individual randomization is adopted. Participants will be recruited over a period of 60 days until the required number has been achieved. The interventions will be administered for a period of 3 months.

Study setting The health facilities for the study will be selected from the Eastern Region. Eastern Region is chosen for the study because it had the highest prevalence of hypertension in 2022 according to the data received from the Ghana Health Service.

According to the 2021 Population and Housing Census (PHC), Eastern region has 33 districts and a total population of 2,925,653. About 49 percent of the total population are males whilst the remaining are females(Ghana Statistical Service, 2021). The main ethnic groups in the region are Akan, Ewe, Ga-Adangbe and Guan (Ghana Statistical Service, 2013). The major religious group in the region is Christianity with fewer inhabitants belonging to the Islamic and traditional religions. There are also a few others who do not belong to any religion (Ghana Statistical Service, 2013). Approximately 45 percent of the population aged 12 years and over own a mobile phone and ownership in the region is largely urban(Ghana Statistical Service, 2013).

Study Participants and Recruitment The eligibility criteria for all phases of the study include 1) adult aged 18 years or older 2) diagnosed of hypertension 3) has uncontrolled hypertension (i.e. systolic blood pressure ≥140 mmHg and a diastolic blood pressure ≥ 90mmHg) documented in their records on 2 clinic visits 4) has been prescribed at least one antihypertensive medication for a period of 2 months before the study 5) owns a smart phone or has access to one at all times.

The exclusion criteria for the study include 1) Pregnant women with hypertension or within 3 months postpartum 2) Hypertensive patients with diabetes, liver failure or kidney disease 3) Plans to travel out of the country during the period of the study 4) Participating in another mobile health intervention or medication adherence intervention 5) has a psychiatric disease or mental illness 6) has a visual impairment.

Healthcare professionals measuring the vital signs of all patients during their visit to the hospital for a review will identify potential participants and invite them to participate in the study. Trained research assistants will assess the eligibility of the patients who have agreed to participate in the study. Medication adherence of patients will be assessed using the eight-item Morisky Medication Adherence Scale (MMAS-8) (Morisky et al., 2008). The MMAS-8 tool is chosen because it has high validity and reliability coupled with good specificity and sensitivity (Culig & Leppee, 2014; Laghousi et al., 2021). The first seven (7) items on the scale require a yes or no response whereas the eighth item uses a five-point Likert scale (never/rarely to all the time). The total score ranges from 0 to 8 with a score of <6 indicative of non-adherence.

Participants from selected health facilities who are eligible and consent to participate in the study will be randomized into the control and intervention groups. The intervention group patients will receive either phone calls or videos thrice weekly for a period of 3 months in addition to usual care. The interventions will be administered on days and times convenient for the participants. Thrice weekly has been chosen because a similar study conducted by Bhandari et al. (2022) utilized the same frequency to send text messages and found that it improved adherence to antihypertensive medicines. The participants who will receive the video-based intervention will be given 3 gigabytes of data for the study.

The control group will only receive care as usual for the 3 months. Baseline and post-intervention data will be collected. The baseline data comprises general information (name, telephone number, date and time of interview as well as days and time convenient for them to receive the interventions), socio-demographic characteristics, blood pressure measurement, hypertension knowledge and medication adherence rating based on MMAS-8

ELIGIBILITY:
Inclusion Criteria:

* adult aged 18 years or older
* diagnosed of hypertension
* has uncontrolled hypertension (i.e. systolic blood pressure ≥140 mmHg and a diastolic blood pressure ≥ 90mmHg) documented in their records on 2 clinic visits
* has been prescribed at least one antihypertensive medication for a period of 2 months before the study
* owns a smart phone or has access to one at all times.

Exclusion Criteria:

* Pregnant women with hypertension or within 3 months postpartum
* Hypertensive patients with diabetes, liver failure or kidney disease
* Plans to travel out of the country during the period of the study
* Participating in another mobile health intervention or medication adherence intervention
* has a psychiatric disease or mental illness 6) has a visual impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
change in systolic blood pressure | baseline and 3 months
  The systolic blood pressure at baseline will be compared to the systolic pressure at endline. This will help to determine if the intervention has an effect on the blood pressure
Medication adherence measured using the Morisky Medication Adherence Scale-8(MMAS-8) | baseline and 3 months
  Medication adherence will be measured at baseline and then after administering the intervention. MMAS-8 has eight items on the scale. The first seven (7) items on the scale require a yes or no response whereas the eighth item uses a five-point Likert scale (never/rarely to all the time). The total score ranges from 0 to 8 with a score of <6 indicative of non-adherence. A score between 6 < 8 indicates medium adherence whereas a score of 8 shows high adherence.

SECONDARY OUTCOMES:
Proportion of patients with controlled blood pressure | baseline and 3 months
  The proportion of patients with controlled blood pressure after administration of the intervention would be measured
Acceptability of the intervention | 3 months
  Participants in the intervention groups will answer questions on the acceptability of the interventions received at the end of the study i.e after the interventions have administered. The instrument that will be used is based on the Unified Theory of Acceptance and Use of Technology which has 5 -Likert scale. Higher scores indicates acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Asuming, PhD, Study Director — University of Ghana; Gordon Abekah-Nkrumah, PhD, Study Chair — University of Ghana
Locations (1):
- St Joseph Catholic Hospital, Efiduase, Koforidua, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Data set or information that will be shared include study protocol
Supporting Information: Study Protocol
Time Frame: The study protocol will be available
Access Criteria: The study protocol will be available online to all. The study protocol will be shared through publications.